CLINICAL TRIAL: NCT01913288
Title: Exposure to Biological Maternal Sounds in Extremely Preterm Infants: Effects on Short- and Long-term Outcomes
Brief Title: Effects of Mother's Voice and Heartbeat Sounds on Preterm Newborns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Charles H. Hood Foundation (Other); Peter and Elizabeth C. Tower Foundation (Unknown)
Responsible Party: Principal Investigator, Amir Lahav, Instructor in Pediatrics, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009p000936
Record Dates: First submitted 2013-05-16; First posted 2013-08-01 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Preterm Birth
Keywords: neonatal care, preterm, maternal sounds, auditory stimulation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biological Maternal Sounds (Experimental): Daily Exposure to recorded mother's voice and heartbeat sounds via audio systems installed at the bedside
  Interventions: Other: Biological Maternal Sounds
- Hospital Sounds (Sham Comparator): Exposure to standard hospital sounds; routine care.
  Interventions: Other: Biological Maternal Sounds

INTERVENTIONS:
Other: Biological Maternal Sounds

SUMMARY:
The purpose of this RCT is to learn more about how sounds that we experience in the womb can affect early development in premature infants. The investigators are specifically interested determining whether and what types of maternal sensory stimulation can influence physical growth, brain maturation, respiratory stability and early vocalization during postnatal development. The investigators hypothesize that daily exposure to biological maternal sounds, such as mother's voice and heartbeat, will improve both short-term and long-term developmental in premature infants and will increase their potential to grow into healthy children.

DETAILED DESCRIPTION:
The purpose of this RCT is to learn more about how sounds that we experience in the womb can affect early development in premature infants. The investigators are specifically interested determining whether and what types of maternal auditory stimulation can influence physical growth, brain maturation, respiratory stability (including heart rate, respiratory rate and oxygen saturation levels) as well as early vocalization prior to 40 weeks gestation. The investigators hypothesize that daily exposure to biological maternal sounds, such as mother's voice and heartbeat, will improve both short-term and long-term developmental outcomes in premature infants and will increase their potential to grow into healthy children.

ELIGIBILITY:
Inclusion Criteria:

* Born between 24-36 weeks GA.

Exclusion Criteria:

* Chromosomal or congenital anomalies; congenital infections; > grade II IVH;
* maternal use of tobacco, alcohol, or illicit drugs;
* significant abuse or malnutrition during pregnancy,
* failed ABR.
* No exclusions based on gender or ethnicity.

Ages: 24 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2013-05; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Brain volume (DM^3) | Between 36-40 weeks gestation
  Data will be obtained by an MRI brain scan and will be calculated separately for white matter, grey matter, CSF.
Language and cognitive skills | At 12 and 24 months corrected-age
  Data will be obtained using the MacArthur-Bates Communicative Development Inventories (CDI), the Receptive-Expressive Emergent Language Test Third Edition (REEL-3), and the Bayley Scales of Infant Development Third Edition (Bayley-III).

SECONDARY OUTCOMES:
Oxygen saturation levels (mg/l) | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  Data will be collected from the bedside cardiac monitor
Heart rate (BPM) | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  Data will be collected from the bedside cardiac monitor
Infant vocalization (word count) | Between 32-36 weeks gesation
  Data will be obtained by real-time recording of the language environment
Weight gain (gr/kg/day) | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  Data will be obtained from medical records

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lahav, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States